CLINICAL TRIAL: NCT02490475
Title: A Phase Ib, Open-Label, Multicenter Study of the Safety and Pharmacokinetics of the Combination of RhuMab 2C4 (Omnitarg), a Recombinant Humanized Antibody to HER2, and Docetaxel (Taxotere) in Patients With Advanced Solid Tumors
Brief Title: A Multiple-Dose Study of RhuMab 2C4 and Docetaxel in the Treatment of Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO17021
Record Dates: First submitted 2015-07-02; First posted 2015-07-03 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Docetaxel; pertuzumab

ARMS (3):
- RhuMab 2C4 + Docetaxel 100 mg/m^2 (Level 3) (Experimental): Docetaxel will be administered via intravenous (IV) infusion on Day 1 of each 3-week cycle at a dose of 100 mg/m^2 per day, and rhuMab 2C4 will be given on Day 1 of each 3-week cycle as a fixed-dose 420-mg IV infusion. For Cycle 1 only, rhuMab 2C4 administration will be delayed to Day 2 with an initial 840-mg loading dose. The incidence of DLTs will be used to guide intrapatient dose modification, as well as subsequent enrollment.
  Interventions: Drug: Docetaxel; Drug: RhuMab 2C4
- RhuMab 2C4 + Docetaxel 60 mg/m^2 (Level 1) (Experimental): Docetaxel will be administered via IV infusion on Day 1 of each 3-week cycle at a dose of 60 mg/m^2 per day, and rhuMab 2C4 will be given on Day 1 of each 3-week cycle as a fixed-dose 420-mg IV infusion. For Cycle 1 only, rhuMab 2C4 administration will be delayed to Day 2 with an initial 840-mg loading dose. The incidence of DLTs will be used to guide intrapatient dose modification, as well as subsequent enrollment.
  Interventions: Drug: Docetaxel; Drug: RhuMab 2C4
- RhuMab 2C4 + Docetaxel 75 mg/m^2 (Level 2) (Experimental): Docetaxel will be administered via IV infusion on Day 1 of each 3-week cycle at a dose of 75 mg/m^2 per day, and rhuMab 2C4 will be given on Day 1 of each 3-week cycle as a fixed-dose 420-mg IV infusion. For Cycle 1 only, rhuMab 2C4 administration will be delayed to Day 2 with an initial 840-mg loading dose. The incidence of DLTs will be used to guide intrapatient dose modification, as well as subsequent enrollment.
  Interventions: Drug: Docetaxel; Drug: RhuMab 2C4

INTERVENTIONS:
Drug: Docetaxel — Participants will receive docetaxel on Day 1 of each 3-week cycle as 60, 75, or 100 mg/m^2 via IV infusion. Treatment may continue until disease progression, unacceptable toxicity, or consent withdrawal.
  Other Names: Taxotere
Drug: RhuMab 2C4 — Participants will receive rhuMab 2C4 on Day 1 of each 3-week cycle as 420 mg via IV infusion. For Cycle 1 ony, rhuMab will be administered on Day 2, at least 24 hours after docetaxel and following an initial 840-mg loading dose. Treatment may continue until disease progression, unacceptable toxicity, or consent withdrawal.
  Other Names: Omnitarg

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics of the combination of rhuMab 2C4 (Perjeta) and docetaxel (Taxotere) in participants with advanced solid tumors that have progressed during or after standard therapy, or for which no standard therapy is available. Participants will be enrolled and evaluated for dose-limiting toxicities (DLTs) in escalating-dose cohorts in order to determine the maximum tolerated dose (MTD).

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age
* Easter Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy at least 12 weeks
* Locally advanced or metastatic solid tumor with at least 1 measurable lesion, which has progressed during/after standard therapy
* Human epidermal growth factor receptor 2 (HER2)-negative among participants with breast cancer
* Negative pregnancy test or use of an adequate contraceptive method among women of childbearing potential
* Adequate hematologic, hepatic, and renal function
* Signed informed consent, histologically or cytologicall confirmed advanced solid tumor, adequate cardiac function as documented by LVEF >50% by ECHO or MUGA

Exclusion Criteria:

* Clinical evidence of central nervous system (CNS) metastases
* Prior chemotherapy, radiotherapy, or immunotherapy within 4 weeks, or hormone therapy within 2 weeks of study Day 1
* History of neuropathy Grade 2 or worse, or any unresolved residual chemotherapy effects
* Prior HER2-active agents or docetaxel
* Any investigational agent within 28 days of study drug
* Prior cumulative doxorubicin dose greater than (>) 360 mg/m^2 or equivalent
* Significant cardiovascular disease
* Active/uncontrolled concurrent illness or infection-
* Major surgery or trauma within 4 weeks of study Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-02; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Rotterdam, Netherlands
- Sutton, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel 60 Plus (+) Pertuzumab 1050: Participants received 60 milligrams per square meter (mg/m^2) docetaxel and 1050 mg of pertuzumab as an intravenous (IV) infusion every 3 weeks until disease progression, unacceptable toxicity, or consent withdrawal. In Cycle 1 docetaxel was administered on Day 1 and pertuzumab was administered at least 24 hours (h) apart on Day 2. Cycle 2 onwards pertuzumab was administered on Day 1 immediately followed by docetaxel. In addition all participants received 8 mg of dexamethasone or its equivalent as corticosteroid premedication.
- Docetaxel 75 + Pertuzumab 1050: Participants received 75 mg/m^2 docetaxel and 1050 mg of pertuzumab as an IV infusion every 3 weeks until disease progression, unacceptable toxicity, or consent withdrawal. In Cycle 1 docetaxel was administered on Day 1 and pertuzumab was administered at least 24 h apart on Day 2. Cycle 2 onwards pertuzumab was administered on Day 1 immediately followed by docetaxel. In addition all participants received 8 mg of dexamethasone or its equivalent as corticosteroid premedication.
- Docetaxel 75 + Pertuzumab 420: Participants received 75 mg/m^2 docetaxel and 420 mg of pertuzumab as an IV infusion every 3 weeks until disease progression, unacceptable toxicity, or consent withdrawal. In Cycle 1 participants received a loading dose of 840 mg of pertuzumab as an IV infusion. Further in Cycle 1 Docetaxel was administered on Day 1 and pertuzumab was administered at least 24 h apart on Day 2. Cycle 2 onwards pertuzumab was administered on Day 1 immediately followed by docetaxel. In addition all participants received 8 mg of dexamethasone or its equivalent as corticosteroid premedication.
- Docetaxel 100 + Pertuzumab 420: Participants received 100 mg/m^2 docetaxel and 420 mg of pertuzumab as an IV infusion every 3 weeks until disease progression, unacceptable toxicity, or consent withdrawal. In Cycle 1 participants received a loading dose of 840 mg of pertuzumab as an IV infusion. Further in Cycle 1 Docetaxel was administered on Day 1 and pertuzumab was administered at least 24 h apart on Day 2. Cycle 2 onwards pertuzumab was administered on Day 1 immediately followed by docetaxel. In addition all participants received 8 mg of dexamethasone or its equivalent as corticosteroid premedication.
Period: Period 1: First 6 Cycles
Arm/Group | Docetaxel 60 Plus (+) Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 420 | Docetaxel 100 + Pertuzumab 420
Started | 6 | 2 | 6 | 5
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 2 | 6 | 5
Not completed — Adverse Event | 2 | 1 | 0 | 1
Not completed — Insufficient Therapeutic Response | 2 | 0 | 2 | 2
Not completed — Refused Treatment | 1 | 0 | 0 | 0
Not completed — Completed 6 Cycles of Therapy | 1 | 1 | 4 | 2
Period: Period 2: Extension Phase
Arm/Group | Docetaxel 60 Plus (+) Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 420 | Docetaxel 100 + Pertuzumab 420
Started | 1 | 0 | 3 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 3 | 1
Not completed — Insufficient Therapeutic Response | 1 | 0 | 2 | 0
Not completed — Refused Treatment | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-To-Treat (ITT) Population included all participants who received any amount of the study medication.
Groups:
- Docetaxel 60 Plus (+) Pertuzumab 1050: Participants received 60 mg/m^2 docetaxel and 1050 mg of pertuzumab as an IV infusion every 3 weeks until disease progression, unacceptable toxicity, or consent withdrawal. In Cycle 1 docetaxel was administered on Day 1 and pertuzumab was administered at least 24 h apart on Day 2. Cycle 2 onwards pertuzumab was administered on Day 1 immediately followed by docetaxel. In addition all participants received 8 mg of dexamethasone or its equivalent as corticosteroid premedication.
- Total: Total of all reporting groups
Arm/Group | Docetaxel 60 Plus (+) Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 420 | Docetaxel 100 + Pertuzumab 420 | Total
Number analyzed (Participants) | 6 | 2 | 6 | 5 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (5.38) | 62.5 (9.19) | 59.5 (6.06) | 45.0 (20.21) | 55.6 (12.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 1 | 3 | 6
  Male | 4 | 2 | 5 | 2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Docetaxel in Combination of Pertuzumab
Description: A prior dose level was defined as an MTD if at a certain dose level, there were greater than or equal to (≥) 2 out of 6 participants who had Dose Limiting Toxicities (DLTs). If there were no DLTs or DLTs were seen in less than (<) 2 participants in the highest dose level, that was considered as MTD. Participants received escalating doses of docetaxel and pertuzumab until DLTs were observed. DLTs were defined as any of the following: 1) Any non-hematological toxicity ≥ Grade 3 according to Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 except for fever, chills and flu-like symptoms, in spite of adequate toxicity management, 2) Grade 4 neutropenia lasting greater than (>) 7 days, 3) Febrile neutropenia, 4) Thrombocytopenia Grade 4 or any thrombocytopenia requiring platelet transfusion or 5) Any subjectively intolerable toxicity felt by the investigator to be related to either one of the compounds.
Time Frame: Cycle 1 Up to Day 15
Population: Safety Population: included all participants who received any amount of study medication and who had at least one post-baseline safety follow-up.
Measure: Number; unit: mg/m^2
Groups:
- Entire Study Population: Participants received escalating dose levels of combination of docetaxel and pertuzumab. Participants received docetaxel 60 mg/m^2 and pertuzumab 1050 mg at dose level 1, docetaxel 75 mg/m^2 and pertuzumab 1050 mg at dose level 2, docetaxel 75 mg/m^2 and pertuzumab 420 mg at dose level 3 or 100 mg/m^2 and pertuzumab 420 mg at dose level 4 until DLTs were observed.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 19
mg/m^2 | 75.0

2. Secondary Outcome: Plasma Decay Half Life (t1/2) for Pertuzumab in Combination With Docetaxel
Description: The biological half-life or terminal half-life of pertuzumab is the time in days it takes for it to lose half of its pharmacologic activity.
Time Frame: Cycle1: Day 2 Pre-dose and 15 minutes, 1.5, 4 and 8 hours Post-dose, and Days 3, 6, 9 and 16; Cycle 2: Day 1 Pre-dose and 15 minutes Post-dose on Days 1, 8, 15 and 22
Population: ITT population; Participants in any cohort infused with the specified dose of pertuzumab were included in analysis. number (n) equals (=) number of participants analyzed at the specified timepoint for each arm, respectively.
Measure: Median (Full Range); unit: days
Groups:
- Pertuzumab 1050: Participants received 1050 mg of pertuzumab in Cycle 1 Day 2 (24 h after the administration of docetaxel) as an IV infusion over approximately 90 minutes and in Cycle 2 on Day 1, (immediately before docetaxel) infused over 30 minutes.
- Pertuzumab 840; Pertuzumab 420: Participants received pertuzumab 840 mg by IV infusion over approximately 90 minutes in Cycle 1 followed by a three weekly dose (Cycle 2) of 420 mg by IV infusion over approximately 30 minutes.
Arm/Group | Pertuzumab 1050 | Pertuzumab 840 | Pertuzumab 420
Number analyzed (Participants) | 8 | 11 | 10
days
  Cycle 1 (n=8,11,0) | 12.65 [7.80 to 19.59] | 11.65 [6.95 to 25.96] | NA [NA to NA] — Participants received 420 mg of pertuzumab only in Cycle 2 per dose regimen.
  Cycle 2 (n=7,0,10) | 19.02 [9.02 to 49.63] | NA [NA to NA] — Participants received 840 mg of pertuzumab only in Cycle 1 per dose regimen. | 18.46 [8.85 to 42.00]

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Pertuzumab in Combination With Docetaxel
Description: Cmax refers to the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and prior to the administration of a second dose and is measures as micrograms per milliliter (μg/mL).
Time Frame: as for outcome 2
Population: ITT population; Participants in any cohort infused with the specified dose of pertuzumab were included in analysis. n = number of participants analyzed at the specified timepoint for each arm, respectively.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Pertuzumab 1050 | Pertuzumab 840 | Pertuzumab 420
Number analyzed (Participants) | 8 | 11 | 10
μg/mL
  Cycle 1 (n=8,11,0) | 301.0 (93.0) | 255.0 (84.0) | NA (NA) — Participants received 420 mg of pertuzumab only in Cycle 2 per dose regimen.
  Cycle 2 (n=7,0,10) | 368.0 (79.0) | NA (NA) — Participants received 840 mg of pertuzumab only in Cycle 1 per dose regimen. | 150.0 (43.0)

4. Secondary Outcome: Area Under the Concentration Curve From Time Zero to the Last Visit (AUC [0-last]) for Pertuzumab in Combination With Docetaxel
Description: The area under the plot of plasma concentration of drug against time after drug administration is defined as the area under the curve (AUC). The AUC0-last is calculated from time 0 (prior to administration of medication) to last measured data point. The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. AUC is measured as micrograms times days per milliliter (μg*day/mL).
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Pertuzumab 1050 | Pertuzumab 840 | Pertuzumab 420
Number analyzed (Participants) | 8 | 11 | 10
μg*day/mL
  Cycle 1 (n=8,11,0) | 2390 (584) | 1749 (543) | NA (NA) — Participants received 420 mg of pertuzumab only in Cycle 2 per dose regimen.
  Cycle 2 (n=7,0,10) | 3500 (551) | NA (NA) — Participants received 840 mg of pertuzumab only in Cycle 1 per dose regimen. | 1491 (472)

5. Secondary Outcome: AUC From Time Zero to Infinity (AUC [0-infinity]) for Pertuzumab in Combination With Docetaxel
Description: The AUC0-infinity is calculated from time 0 (prior to administration of medication) to infinity (the time of complete elimination of the drug). The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. AUC is measured as μg*day/mL.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μg*day/mL
Arm/Group | Pertuzumab 1050 | Pertuzumab 840 | Pertuzumab 420
Number analyzed (Participants) | 8 | 11 | 10
μg*day/mL
  Cycle 1 (n=8,11,0) | 3951 (919) | 2796 (967) | NA (NA) — Participants received 420 mg of pertuzumab only in Cycle 2 per dose regimen
  Cycle 2 (n=7,0,10) | 6856 (2335) | NA (NA) — Participants received 840 mg of pertuzumab only in Cycle 1 per dose regimen. | 2762 (892)

6. Secondary Outcome: Clearance (Cl) of Pertuzimab in Combination With Docetaxel
Description: Clearance (expressed as volume/time) describes the removal of drug from a volume of plasma in a given unit of time (drug loss from the body). It is measured as milliliters per day (mL/day).
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | Pertuzumab 1050 | Pertuzumab 840 | Pertuzumab 420
Number analyzed (Participants) | 8 | 11 | 10
mL/day
  Cycle 1 (n=8,11,0) | 282 (83) | 329 (97) | NA (NA) — Participants received 420 mg of pertuzumab only in Cycle 2 per dose regimen.
  Cycle 2 (n=7,0,10) | 167 (49) | NA (NA) — Participants received 840 mg of pertuzumab only in Cycle 1 per dose regimen. | 169 (60)

7. Secondary Outcome: Volume of Distribution (Vz) at Steady State of Pertuzumab in Combination With Docetaxel
Description: The volume of distribution at steady state (Vz), also known as apparent volume of distribution, is a pharmacological, theoretical volume that the total amount of administered drug would have to occupy (if it were uniformly distributed), to provide the same concentration as it currently is in blood plasma.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Pertuzumab 1050 | Pertuzumab 840 | Pertuzumab 420
Number analyzed (Participants) | 8 | 11 | 10
mL
  Cycle 1 (n=8,11,0) | 5214 (1386) | 5355 (1680) | NA (NA) — Participants received 420 mg of pertuzumab only in Cycle 2 per dose regimen.
  Cycle 2 (n=7,0,10) | 4672 (1221) | NA (NA) — Participants received 840 mg of pertuzumab only in Cycle 1 per dose regimen. | 4233 (1555)

8. Secondary Outcome: Mean Residence Time (MRT) of Pertuzumab
Description: MRT is the average time that pertuzumab is present in the systemic circulation and is measured in days.
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Pertuzumab 1050 | Pertuzumab 840 | Pertuzumab 420
Number analyzed (Participants) | 8 | 11 | 10
days
  Cycle 1 (n=8,11,0) | 17.8 (5.8) | 15.8 (6.7) | NA (NA) — Participants received 420 mg of pertuzumab only in Cycle 2 per dose regimen.
  Cycle 2 (n=7,0,10) | 29.5 (18.5) | NA (NA) — Participants received 840 mg of pertuzumab only in Cycle 1 per dose regimen. | 25.8 (13.2)

9. Secondary Outcome: Percentage of Participants by Best Overall Response Using Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Best Overall response was evaluated as Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD). CR: complete disappearance of all target lesions. PR: at least a 30 percent (%) decrease in the sum of the longest diameters. SD: neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum of the longest diameters since the treatment started. PD: at least a 20% increase in the sum of the longest diameters of target lesions, taking as reference the smallest sum of the longest diameters of the target lesions recorded since the treatment started, including screening, or the appearance of one or more new lesions. If participants withdrew due to insufficient therapeutic response or death and had no tumor measurements at the final visit, they were counted under progressive disease for final visit.
Time Frame: Weeks 7 (Cycle 2),13 (Cycle 4) and Final Visit Up to 22 weeks
Population: ITT population; n = number of participants still receiving treatment at the specified cycle for each arm respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel 60 Plus (+) Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 420 | Docetaxel 100 + Pertuzumab 420
Number analyzed (Participants) | 6 | 2 | 6 | 5
percentage of participants
  Cycle 2: CR (n=6,1,6,4) | 0.0 | 0.0 | 0.0 | 0.0
  Cycle 2:PR (n=6,1,6,4) | 0.0 | 0.0 | 0.0 | 0.0
  Cycle 2:SD (n=6,1,6,4) | 83.3 | 100.0 | 83.3 | 75.0
  Cycle 2:PD (n=6,1,6,4) | 16.7 | 0 | 16.7 | 25.0
  Cycle 2:Missing (n=6,1,6,4) | 0.0 | 0.0 | 0.0 | 0.0
  Cycle 4:CR (n=5,1,5,3) | 0.0 | 0.0 | 0.0 | 0.0
  Cycle 4:PR (n=5,1,5,3) | 0.0 | 0.0 | 20.0 | 0
  Cycle 4:SD (n=5,1,5,3) | 80.0 | 100.0 | 40.0 | 66.7
  Cycle 4:PD (n=5,1,5,3) | 20.0 | 0.0 | 40.0 | 33.3
  Cycle 4:Missing (n=5,1,5,3) | 0.0 | 0.0 | 0.0 | 0.0
  Final visit:CR (n=6,2,6,5) | 0.0 | 0.0 | 0.0 | 0.0
  Final visit:PR (n=6,2,6,5) | 0.0 | 0.0 | 16.7 | 0.0
  Final visit:SD (n=6,2,6,5) | 33.3 | 50.0 | 33.3 | 20.0
  Final visit:PD (n=6,2,6,5) | 50.0 | 0.0 | 50.0 | 60.0
  Final visit:Missing (n=6,2,6,5) | 16.7 | 50.0 | 0.0 | 20.0

10. Secondary Outcome: Percentage of Participants With Decrease in Left Ventricular Ejection Fraction (LVEF) by Category of Decrease and Timepoint
Description: Ejection fraction (EF) is the fraction of outbound blood pumped from the heart with each heartbeat. It is commonly measured by echocardiogram and serves as a general measure of a person's cardiac function. Changes in LVEF were assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 criteria. The decrease in LVEF has been categorized as follows: A) Increase, no change, decrease from baseline less than (<) 10%; B) Absolute value <50% and decrease from baseline greater than or equal to (≥) 10%; C) Absolute value <50% and decrease from baseline≥15% ; D) Other. If participants withdrew due to insufficient therapeutic response or death and had no tumor measurements at the final visit, they were counted under progressive disease for final visit.
Time Frame: Baseline, Weeks 7(Cycle 2), 13 (Cycle 4) and Final Visit Up to Week 22
Population: ITT population; n = number of participants still receiving treatment at the specified cycle for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | Docetaxel 60 Plus (+) Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 420 | Docetaxel 100 + Pertuzumab 420
Number analyzed (Participants) | 6 | 2 | 6 | 5
percentage of participants
  Cycle 2: A (n=6,1,6,4) | 83.3 | 100.0 | 100.0 | 100.0
  Cycle 2: B (n=6,1,6,4) | 0.0 | 0.0 | 0.0 | 0.0
  Cycle 2: C (n=6,1,6,4) | 0.0 | 0.0 | 0.0 | 0.0
  Cycle 2: D (n=6,1,6,4) | 16.7 | 0.0 | 0.0 | 0.0
  Cycle 4: A (n=5,1,4,3) | 100.0 | 100.0 | 75.0 | 100.0
  Cycle 4: B (n=5,1,4,3) | 0.0 | 0.0 | 25.0 | 0.0
  Cycle 4: C (n=5,1,4,3) | 0.0 | 0.0 | 0.0 | 0.0
  Cycle 4: D (n=5,1,4,3) | 0.0 | 0.0 | 0.0 | 0.0
  Final Visit: A (n=3,1,5,2) | 66.7 | 100.0 | 80.0 | 100.0
  Final Visit: B (n=3,1,5,2) | 0.0 | 0.0 | 0.0 | 0.0
  Final Visit: C (n=3,1,5,2) | 0.0 | 0.0 | 0.0 | 0.0
  Final Visit: D (n=3,1,5,2) | 33.3 | 0.0 | 20.0 | 0.0

11. Secondary Outcome: t1/2 for Docetaxel Alone and in Combination With Pertuzumab
Description: The biological half-life or terminal half-life of docetaxel is the time in hours it takes for it to lose half of its pharmacologic activity. Data for "docetaxel alone" arms were analyzed for the timepoints on Day 1 prior to the administration of pertuzumab. The pharmacokinetic parameters were derived by non-compartmental methods using WinNonLin version 5.0.1.
Time Frame: Cycles 1 and 2: Pre-dose, 30 and 55 minutes during dosing, 15 minutes, 30 minutes, 1, 2, 4, 8, and 23 hours Post-dose
Population: ITT population; Data from Cohort 2 (docetaxel 75 mg/m^2 and pertuzumab 1050 mg) were excluded because there were only 2 participant data. It was planned not to report PK data, if less than or equal to 2 participants were analyzed. n= number of participants analyzed at the specified cycle.
Measure: Median (Full Range); unit: days
Groups:
- Docetaxel 60 Alone; Docetaxel 60 + Pertuzumab 1050: Participants received 60 mg/m^2 docetaxel and 1050 mg of pertuzumab as an IV infusion every 3 weeks until disease progression, unacceptable toxicity, or consent withdrawal. In Cycle 1 docetaxel was administered on Day 1 and pertuzumab was administered at least 24 h apart on Day 2. Cycle 2 onwards pertuzumab was administered on Day 1 immediately followed by docetaxel. In addition all participants received 8 mg of dexamethasone or its equivalent as corticosteroid premedication.
- Docetaxel 75 Alone; Docetaxel 75+ Pertuzumab 420: Participants received 75 mg/m^2 docetaxel and 420 mg of pertuzumab as an IV infusion every 3 weeks until disease progression, unacceptable toxicity, or consent withdrawal. In Cycle 1 participants received a loading dose of 840 mg of pertuzumab as an IV infusion. Further in Cycle 1 Docetaxel was administered on Day 1 and pertuzumab was administered at least 24 h apart on Day 2. Cycle 2 onwards pertuzumab was administered on Day 1 immediately followed by docetaxel. In addition all participants received 8 mg of dexamethasone or its equivalent as corticosteroid premedication.
- Docetaxel 100 Alone; Docetaxel 100 + Pertuzumab 420: Participants received 100 mg/m^2 docetaxel and 420 mg of pertuzumab as an IV infusion every 3 weeks until disease progression, unacceptable toxicity, or consent withdrawal. In Cycle 1 participants received a loading dose of 840 mg of pertuzumab as an IV infusion. Further in Cycle 1 Docetaxel was administered on Day 1 and pertuzumab was administered at least 24 h apart on Day 2. Cycle 2 onwards pertuzumab was administered on Day 1 immediately followed by docetaxel. In addition all participants received 8 mg of dexamethasone or its equivalent as corticosteroid premedication.
Arm/Group | Docetaxel 60 Alone | Docetaxel 60 + Pertuzumab 1050 | Docetaxel 75 Alone | Docetaxel 75+ Pertuzumab 420 | Docetaxel 100 Alone | Docetaxel 100 + Pertuzumab 420
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 4
days
  Cycle 1 (n=6,0,6,0,5,0) | 17.7 [7.31 to 22.7] | NA [NA to NA] — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only. | 12.0 [9.56 to 19.4] | NA [NA to NA] — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only. | 8.92 [7.49 to 13.5] | NA [NA to NA] — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only.
  Cycle 2(n=0,6,0,6,0,4) | NA [NA to NA] — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 19.7 [12.5 to 27.1] | NA [NA to NA] — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 13.8 [9.62 to 23.8] | NA [NA to NA] — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 11.8 [8.04 to 21.4]

12. Secondary Outcome: Tmax for Docetaxel Alone and in Combination With Pertuzumab
Description: Tmax is defined as the time after administration of a drug when the maximum plasma concentration is reached; Data for "docetaxel alone" arms were analyzed for the timepoints on Day 1 prior to the administration of pertuzumab. When the rate of absorption equals the rate of elimination. The pharmacokinetic parameters were derived by non-compartmental methods using WinNonLin version 5.0.1.
Time Frame: Cycles 1 and 2: Pre-dose, 30 and 55 minutes during dosing, 15 minutes, 30 minutes, 1, 2, 4, 8, and 23 hours Post-dose
Population: as for outcome 11
Measure: Median (Full Range); unit: days
Arm/Group | Docetaxel 60 Alone | Docetaxel 60 + Pertuzumab 1050 | Docetaxel 75 Alone | Docetaxel 75 + Pertuzumab 420 | Docetaxel 100 Alone | Docetaxel 100 + Pertuzumab 420
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 4
days
  Cycle 1 (n=6,0,6,0,5,0) | 0.50 [0.50 to 0.90] | NA [NA to NA] — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only. | 0.50 [0.50 to 0.90] | NA [NA to NA] — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only. | 0.90 [0.90 to 0.90] | NA [NA to NA] — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only.
  Cycle 2 (n=0,6,0,6,0,4) | NA [NA to NA] — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 0.90 [0.50 to 1.25] | NA [NA to NA] — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 0.90 [0.50 to 0.90] | NA [NA to NA] — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 0.70 [0.50 to 0.90]

13. Secondary Outcome: Cmax for Docetaxel Alone and in Combination With Pertuzumab
Description: Cmax refers to the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and prior to the administration of a second dose and is measures as nanograms per milliliter (ng/mL). The pharmacokinetic parameters were derived by non-compartmental methods using WinNonLin version 5.0.1.
Time Frame: Cycles 1 and 2: Pre-dose, 30 and 55 minutes during dosing, 15 minutes, 30 minutes, 1, 2, 4, 8, and 23 hours Post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Docetaxel 60 Alone | Docetaxel 60 + Pertuzumab 1050 | Docetaxel 75 Alone | Docetaxel 75 + Pertuzumab 420 | Docetaxel 100 Alone | Docetaxel 100 + Pertuzumab 420
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 4
ng/mL
  Cycle 1 (n=6,0,6,0,5,0) | 1642 (274) | NA (NA) — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only. | 3128 (895) | NA (NA) — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only. | 5450 (1867) | NA (NA) — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only.
  Cycle 2 (n=0,6,0,6,0,4) | NA (NA) — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 1695 (331) | NA (NA) — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 2722 (912) | NA (NA) — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 4705 (1871)

14. Secondary Outcome: AUC(0-∞) for Docetaxel Alone and in Combination With Pertuzumab
Description: The AUC0-infinity is calculated from time 0 (prior to administration of medication) to infinity (the time of complete elimination of the drug). The AUC is of particular use in estimating the bioavailability of drugs, by measuring the extent of absorption. AUC is measured as ng*h/mL. The pharmacokinetic parameters were derived by non-compartmental methods using WinNonLin version 5.0.1.
Time Frame: Cycles 1 and 2: Pre-dose, 30 and 55 minutes during dosing, 15 minutes, 30 minutes, 1, 2, 4, 8, and 23 hours Post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Docetaxel 60 Alone | Docetaxel 60 + Pertuzumab 1050 | Docetaxel 75 Alone | Docetaxel 75 + Pertuzumab 420 | Docetaxel 100 Alone | Docetaxel 100 + Pertuzumab 420
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 4
ng*h/mL
  Cycle 1 (n=6,0,6,0,5,0) | 1838 (244) | NA (NA) — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only. | 3744 (1304) | NA (NA) — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only. | 5930 (2137) | NA (NA) — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only.
  Cycle 2 (n=0,6,0,6,0,4) | NA (NA) — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 1734 (409) | NA (NA) — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 3496 (1211) | NA (NA) — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 5218 (2216)

15. Secondary Outcome: Vss for Docetaxel Alone and in Combination With Pertuzumab
Description: The volume of distribution at steady state (Vss), also known as apparent volume of distribution, is a pharmacological, theoretical volume that the total amount of administered drug would have to occupy (if it were uniformly distributed), to provide the same concentration as it currently is in blood plasma. The pharmacokinetic parameters were derived by non-compartmental methods using WinNonLin version 5.0.1.
Time Frame: Cycles 1 and 2: Pre-dose, 30 and 55 minutes during dosing, 15 minutes, 30 minutes, 1, 2, 4, 8, and 23 hours Post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Docetaxel 60 Alone | Docetaxel 60 + Pertuzumab 1050 | Docetaxel 75 Alone | Docetaxel 75 + Pertuzumab 420 | Docetaxel 100 Alone | Docetaxel 100 + Pertuzumab 420
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 4
mL/m^2
  Cycle 1 (n=6,0,6,0,5,0) | 786981 (218139) | NA (NA) — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only. | 410174 (184216) | NA (NA) — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only. | 254233 (85054) | NA (NA) — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only.
  Cycle 2 (n=0,6,0,6,0,4) | NA (NA) — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 1023569 (335711) | NA (NA) — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 566759 (361946) | NA (NA) — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 428863 (283977)

16. Secondary Outcome: CL for Docetaxel Alone and in Combination With Pertuzumab
Description: Clearance (expressed as volume/time) describes the removal of drug from a volume of plasma in a given unit of time (drug loss from the body). It is measured as milliliters per hour per meter squared (mL/h/m^2). The pharmacokinetic parameters were derived by non-compartmental methods using WinNonLin version 5.0.1.
Time Frame: Cycles 1 and 2: Pre-dose, 30 and 55 minutes during dosing, 15 minutes, 30 minutes, 1, 2, 4, 8, and 23 hours Post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mL/h/m^2
Arm/Group | Docetaxel 60 Alone | Docetaxel 60 + Pertuzumab 1050 | Docetaxel 75 Alone | Docetaxel 75 + Pertuzumab 420 | Docetaxel 100 Alone | Docetaxel 100 + Pertuzumab 420
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 5 | 4
mL/h/m^2
  Cycle 1 (n=6,0,6,0,5,0) | 33128 (4396) | NA (NA) — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only. | 22013 (7031) | NA (NA) — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only. | 18913 (7245) | NA (NA) — In Cycle 1 analysis was performed for docetaxel alone data on pertuzumab naive participants only.
  Cycle 2 (n=0,6,0,6,0,4) | NA (NA) — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 35813 (6216) | NA (NA) — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 23747 (8175) | NA (NA) — Data were not analyzed for docetaxel alone since participants were already exposed to pertuzumab in Cycle 1. | 22976 (12679)

17. Secondary Outcome: Number of Participants With DLTs
Description: DLTs were defined as any of the following: 1) Any non-hematological toxicity greter than or equal to (≥) Grade 3 according t0 CTCAE version 3.0 except for fever, chills and flu-like symptoms, in spite of adequate toxicity management, 2) Grade 4 neutropenia lasting greater than (>) 7 days, 3) Febrile neutropenia, 4) Thrombocytopenia Grade 4 or any thrombocytopenia requiring platelet transfusion or 5) Any subjectively intolerable toxicity felt by the investigator to be related to either one of the compounds.
Time Frame: From Baseline until 4 weeks after the end of treatment
Population: Safety Population
Measure: Number; unit: number of participants
Arm/Group | Docetaxel 60 Plus (+) Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 420 | Docetaxel 100 + Pertuzumab 420
Number analyzed (Participants) | 6 | 2 | 6 | 5
number of participants | 0 | 2 | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were continuously monitored from Screening until 4 weeks after the final visit.
Arm/Group | Docetaxel 60 Plus (+) Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 1050 | Docetaxel 75 + Pertuzumab 420 | Docetaxel 100 + Pertuzumab 420
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/2 | 0/6 | 3/5
Other Adverse Events (participants affected / at risk) | 6/6 | 2/2 | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel 60 Plus (+) Pertuzumab 1050 (N=6) | Docetaxel 75 + Pertuzumab 1050 (N=2) | Docetaxel 75 + Pertuzumab 420 (N=6) | Docetaxel 100 + Pertuzumab 420 (N=5)
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel 60 Plus (+) Pertuzumab 1050 (N=6) | Docetaxel 75 + Pertuzumab 1050 (N=2) | Docetaxel 75 + Pertuzumab 420 (N=6) | Docetaxel 100 + Pertuzumab 420 (N=5)
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 5 | 4
Nausea (Gastrointestinal disorders) | 5 | 2 | 5 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 3 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 5 | 2 | 6 | 5
Mucosal inflammation (General disorders) | 2 | 0 | 2 | 1
Malaise (General disorders) | 2 | 0 | 1 | 1
Oedema peripheral (General disorders) | 1 | 0 | 1 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 2
Extravasation (General disorders) | 1 | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Suprapubic pain (General disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 1 | 4 | 0
Headache (Nervous system disorders) | 1 | 0 | 2 | 2
Paraesthesia (Nervous system disorders) | 1 | 0 | 1 | 0
Ageusia (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 4 | 0 | 2 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 1
Lacrimation (Eye disorders) | 1 | 0 | 2 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ventricular disfunction (Cardiac disorders) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Gential Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.